CLINICAL TRIAL: NCT02313818
Title: Variable-length Cognitive Processing Therapy for Combat-Related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Boston VA Research Institute, Inc. (Other); The University of Texas Health Science Center at San Antonio (Other); STRONG STAR Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062853; W81XWH-13-2-0012 (Other: VA Boston Healthcare System)
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Cognitive Processing Therapy; Active Duty Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Variable length Cognitive Processing Therapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPT-C (Experimental): Cognitive Processing Therapy-Cognitive Only (CPT-C) conducted twice weekly for 4-24 sessions based on good end state functioning.
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive Only

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy-Cognitive Only — Cognitive Processing Therapy-Cognitive Only (CPT-C) is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Individual sessions will be conducted twice weekly for 4-24 sessions; each session is 60 minutes.

SUMMARY:
The primary goal of this study is to improve the overall efficacy of cognitive processing therapy-cognitive-only version (CPT-C) in a sample of 130 active-duty service members through a variable length treatment.

DETAILED DESCRIPTION:
The primary goal of this study is to improve the overall efficacy of cognitive processing therapy-cognitive-only version (CPT-C) in a sample of 130 active-duty service members through a variable length treatment. The study seeks to determine if some service members would benefit from a longer or shorter dose of treatment (4-24 sessions), and to identify which individuals are likely to require more, less, or the standard number of treatment sessions to reach good end-state functioning. Predictors of length of therapy and treatment outcome will be examined. Specifically, we will evaluate factors related to internalizing/externalizing traits, cognitive flexibility, inability to inhibit dysfunctional cognitions, and readiness to change as they are related to the number of treatment sessions required to treat patients to the point of good end-state functioning. Additional outcomes including alcohol use, psychosocial functioning, physical health, and sleep also will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female combat veterans who deployed in support of combat operations following 9/11
* Diagnosis of PTSD determined by a Clinician-Administered Posttraumatic Stress Scale (CAPS-5)
* Speak and read English

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention.
* Active psychosis.
* Moderate to severe brain damage (as determined by the inability to comprehend the baseline screening questionnaires).
* Local availability of fewer than 5 months
* Late-phase Med Board status, awaiting percentages
* Undergoing a chapter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PTSD symptoms as measured by thePosttraumatic Stress Disorder Checklist-5 (PCL-5) | Pretreatment, weekly during treatment, 4 weeks, 12 weeks, and 24 weeks posttreatment
  PCL-5 measures symptoms of posttraumatic stress disorder in response to a specific stressor.
Change from baseline in PTSD symptoms as measured by the Clinician Administered PTSD Scale (CAPS-5) | Pretreatment, weekly during treatment, 4 weeks, 12 weeks, and 24 weeks posttreatment
  is an updated version of the gold standard CAPS designed to assess the criteria for PTSD as defined by the DSM-5

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms as measured by the Patient Health Questionnaire-9 | Pretreatment, weekly during treatment, 4 weeks, 12 weeks, and 24 weeks posttreatment
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms (Kroenke, Spitzer, & Williams, 2001). It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the diagnostic criteria for DSM MDD. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed to obtain a total severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Resick, PhD, Principal Investigator — Duke University
Locations (1):
- Carl R Darnall Army Medical Center, Fort Hood, Texas, United States

REFERENCES:
- [Derived] Hass NC, Wachen JS, Straud CL, Checko E, McGeary DD, McGeary CA, Mintz J, Litz BT, Young-McCaughan S, Yarvis JS, Peterson AL, Resick PA; STRONG STAR Consortium. Changes in pain and related health outcomes after cognitive processing therapy in an active duty military sample. J Trauma Stress. 2025 Jun;38(3):447-457. doi: 10.1002/jts.23143. Epub 2025 Mar 5. PMID 40045687
- [Derived] Foa EB, Zandberg LJ, McLean CP, Rosenfield D, Fitzgerald H, Tuerk PW, Wangelin BC, Young-McCaughan S, Peterson AL. The efficacy of 90-minute versus 60-minute sessions of prolonged exposure for posttraumatic stress disorder: Design of a randomized controlled trial in active duty military personnel. Psychol Trauma. 2019 Mar;11(3):307-313. doi: 10.1037/tra0000351. Epub 2018 Feb 12. PMID 29431455